CLINICAL TRIAL: NCT05106660
Title: Safety and Efficacy of Same Day vs Next Day Discharge Post Sleeve Gastrectomy
Brief Title: Ambulatory Laparoscopic Sleeve Gastrectomy
Acronym: DAYSLEEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: New You Medical Center (Unknown)
Responsible Party: Principal Investigator, Aayed Alqahtani, Professor of Surgery, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYASCLSG001
Record Dates: First submitted 2021-10-13; First posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Obesity, Morbid
Keywords: sleeve gastrectomy; ambulatory surgery; day case surgery
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambulatory Care Laparoscopic sleeve gastrectomy (Experimental): Laparoscopic sleeve gastrectomy as ambulatory care procedure with same-day discharge
  Interventions: Procedure: Ambulatory Laparoscopic Sleeve Gastrectomy
- Next Day Discharge Laparoscopic sleeve gastrectomy (Active Comparator): Laparoscopic sleeve gastrectomy with next day discharge
  Interventions: Procedure: Conventional Laparoscopic Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Ambulatory Laparoscopic Sleeve Gastrectomy — Same-day discharge
  Arms: Ambulatory Care Laparoscopic sleeve gastrectomy
Procedure: Conventional Laparoscopic Sleeve Gastrectomy — Next-day discharge
  Arms: Next Day Discharge Laparoscopic sleeve gastrectomy

SUMMARY:
In the era of laparoscopic surgery, day case procedures are increasingly practiced around the world, however, day case bariatric surgery remains a controversial issue due to lack of sufficient evidence evaluating its safety. Laparoscopic sleeve gastrectomy (LSG) is currently the most popular bariatric surgery performed worldwide, and the standard is 1-2 days postop stay. However, the American College of Surgeons and the American Society for Metabolic and Bariatric Surgery released guidelines in 2016 that allowed LSG in ambulatory surgery centers for low acuity patients. In the present trial, investigators will compare the safety and feasibility of same day discharge vs next day discharge in a large group of patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
This is a 2-group, randomized, open label clinical trial patients who will be recruited at an ASC to undergo LSG with same-day discharge, termed Ambulatory Surgery Center LSG (ASC LSG) or LSG with conventional hospitalization and next day discharge (CH LSG). The study will recruit participants between December 2018 and December 2020. Data collected will include including age, body mass index (BMI), operative time, recovery room time, hospital stay, readmission, follow up visits, ASC visits, adverse events, and re-operation rates.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years
2. Body mass index <60
3. American Anesthesiologists Association classification ≤III
4. Commitment to stay within close proximity to the ambulatory surgery center for 4 days after surgery

Exclusion Criteria:

1. High risk for thromboembolic disease
2. Has a history of major open abdominal surgery
3. Bleeding disorders
4. Heart disease
5. Pulmonary hypertension
6. Uncontrolled type 2 diabetes
7. Severe obstructive sleep apnea
8. Chronic obstructive pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Readmission | up to 12 months after surgery
  Readmission to hospital after discharge
Number of patients undergoing reoperative or revisional surgical or endoscopic intervention | up to 12 months
  Number of participants who underwent abdominal surgery or endoscopy for sleeve gastrectomy related complications
Hospital Transfer | up to 16 hours
  Transfer of patient in Ambulatory LSG group to hospital for postop stay
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | within 30 days
  Number of participants who experienced postoperative complications (e.g. bleeding, staple line leaks, surgical site infection, etc...)
Mortality | up to 30 days
  Postoperative 30-day mortality rate

SECONDARY OUTCOMES:
Weight loss | 3 months, 6 months, and 1 year
  Weight difference between baseline and follow-up visits in kilograms. Weight measured using validated, calibrated scale with minimal clothing.

CONTACTS AND LOCATIONS:
Overall Officials: Aayed Alqahtani, MD FRCSC, Principal Investigator — New You Medical Center
Locations (1):
- New You Medical Center, Riyadh, Saudi Arabia